CLINICAL TRIAL: NCT04690894
Title: Ultrasound-guided Erector Spinae Muscle Block Versus Ultrasound-guided Caudal Block in Pediatric Patient Undergoing Lower Abdominal Surgery
Brief Title: Erector Spinae Muscle Block Versus Caudal Block by Sonar in Pediatrics Undergoing Lower Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Shadwa Rabea Mohamed, lecturer, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 266:7/2019
Record Dates: First submitted 2020-12-28; First posted 2020-12-31 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2019-05

CONDITIONS: Postoperative Analgesia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Erector spinae group (Active Comparator): the child received ultrasound-guided erector spinae muscle block in a dose of 0.4mg/kg of 0.25%bupivacaine between the 10th transverse process and erector spinae muscle
  Interventions: Procedure: erector spinae block - caudal block
- caudal group (Active Comparator): child received ultrasound-guided caudal block in a dose of 2.5mg/kg of bupivacaine 0.25%
  Interventions: Procedure: erector spinae block - caudal block
- control (No Intervention): child didn't received any regional block

INTERVENTIONS:
Procedure: erector spinae block - caudal block — the child placed in lateral position identification of spinous process of 10th thoracic vertebral then the transducer was moved 2.5 cm laterally to visualize the transverse process and a total of 0.4mg/kg of 0.25%bupivacaine was adminstered
  Arms: Erector spinae group; caudal group

SUMMARY:
this prospective randomized double blind controlled study was conducted on 60 child scheduled for lower abdominal surgery under general anesthesia. the patients were randomly allocated into 3 parallel groups.group (ESB) patients received ultrasound-guided erector spinae block in a dose of 0.4mg/ml of 0.25%bupivacaine between the 10th transverse process and erector spinae muscles.group(CB) patients received ultrasound-guided caudal block in a dose of 2.5mg/kg of 0.25%bupivacaine. group(CO) did,t received any block

DETAILED DESCRIPTION:
on arrival of the patients to the operative theatre and after placement of the standard monitoring general inhalational anesthesia was induced by face mask with sevoflurane (4-8%) in oxygen after IV cannula was secured patients received 1mic/kg fentanyl and intubation was facilitated by 0.5mg/kg atracurium. isoflurane 1-2% with oxygen was used for maintenance of anesthesia. after stabilization of the patient's hemodynamics and before skin incision erector spinae block or caudal block was performed with the patient in lateral position. after the block patients were flipped back to their normal supine position, surgery took place 10 min after injection of local anesthetic. after termination of surgery reversal of the atracurium was done by giving neostigmine in a dose of 0.04mg/kg and atropine 0.02mg/kg and awake extubation was done

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients aged 2-6 years scheduled for lower abdominal surgery under general anesthesia

Exclusion Criteria:

* parent refusal
* spinal and meningeal anomalies
* mental retardation
* blood disease
* infection at site of injection
* drug allergy

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
number of patients need rescue analgesia | 24 hours
  total number of patients need addition of anagesia

SECONDARY OUTCOMES:
First analgesic request | 24 hours
  First time that patient require analgesia
Hemodynamic changes in the study period | 24 hours
  Changes in HR and blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Talaat, MD, Study Director — professor
Locations (1):
- Faculty of Medicine, Minya, Egypt

REFERENCES:
- [Derived] Abdelrazik AN, Ibrahim IT, Farghaly AE, Mohamed SR. Ultrasound-guided Erector Spinae Muscle Block Versus Ultrasound-guided Caudal Block in Pediatric Patients Undergoing Lower Abdominal Surgeries. Pain Physician. 2022 Jul;25(4):E571-E580. PMID 35793181